CLINICAL TRIAL: NCT04628221
Title: A Single-Arm, Open Label Clinical Study to Collect Safety Data on the Osteoprobe System When Used as a Measurement Tool
Brief Title: Open Label Study Using OsteoProbe System
Acronym: OP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Active Life Scientific, Inc. (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OP2020
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Adverse Effects in the Use of the OsteoProbe System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: OsteoProbe System — The OsteoProbe® System ("OsteoProbe") is a bone microindentation measurement tool. The device is a measurement tool that is not intended to make a diagnosis or provide a treatment decision. There are no other available measurement tools for clinical assessment of bone's resistance to microindentation.

SUMMARY:
Prospective, Single Center, Open Label Clinical Study. The purpose of the study is to collect safety data associated with the use of the OsteoProbe System. Study Duration is expected to take approximately 3 months from first subject enrolled to the last follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Be greater than or equal to 22 years of age;
2. Be able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study
3. If female and of child-bearing potential, must have a negative pregnancy status.

Exclusion Criteria:

1. Active skin infection at the procedure site as identified during a SOC physical examination.
2. Subject-reported or known systemic infection;
3. Subject-reported or known allergy to local anesthetic;
4. Subject-reported or known allergy to stainless steel or nickel materials;
5. Subject-reported or known current use of systemic antibiotics, or topical antibiotics administered to the procedure site;
6. Subject-reported or known history of needle phobia;
7. Significant soft tissue at the procedure site which would preclude use of the OsteoProbe in the judgement of the Investigator;
8. Known instance of hardware in the tibia that is intended to be measured based on radiographic imaging;
9. Known instance of a previous or current fracture in the tibia that is intended to be measured based on radiographic imaging;
10. Are known to be actively participating or known to have participated in another clinical investigation for which they received an investigational product (including but not limited to a drug or vaccine) within the last 90 days, or reports that they intend to participate in another clinical investigation during the course of the study;
11. Are known to be currently abusing drugs or alcohol or have a known history of the same within the last 12 months;
12. Have any known or subject reported mental or psychological disorders that, in the judgement of the Investigator, would impair their ability to accurately complete the NRS Pain Score surveys;
13. Are currently a prisoner;
14. Have a condition which, in the judgement of the Investigator, would preclude adequate evaluation of the device's safety and performance. Conditions include but are not limited to:

    1. Regional or systemic pain syndromes
    2. Radicular pain syndromes
    3. Chronic or intermittent leg pain
    4. Migraine headaches

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Meridian Clinical Research, LLC., Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OsteoProbe System
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.95 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Reported Device Related Serious Adverse Events.
Description: The number of participants who experienced device-related serious adverse events (SAEs) in subjects evaluated with the OsteoProbe System, per potential risks in the protocol.
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
Participants | 0

2. Primary Outcome: The Number of Participants With Reported Device Related Serious Adverse Events.
Description: The incidence of device-related serious adverse events (SAEs) in subjects evaluated with the OsteoProbe System.
Time Frame: 1-day follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
Participants | 0

3. Primary Outcome: The Number of Participants With Reported Device Related Serious Adverse Events.
Description: The incidence of device-related serious adverse events (SAEs) in subjects evaluated with the OsteoProbe System.
Time Frame: 7-day follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
Participants | 0

4. Primary Outcome: The Number of Participants With Reported Device Related Serious Adverse Events.
Description: as for outcome 1
Time Frame: 30-day follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
Participants | 0

5. Secondary Outcome: NRS Pain Scores
Description: The Numeric Rating Scale (NRS) is a continuous scale comprised of a line, with an eleven point numeric range (0 to 10) anchored by 2 verbal descriptors, one for each symptom extreme. The 0 mark corresponds to 'no pain', while the 10 mark corresponds to 'worse pain possible'. Therefore, higher scores indicate greater pain intensity. At all follow-up time points (post-procedure, Day 1, Day 7 , and Day 30), average was taken compared to baseline (Pre-Procedure).
Time Frame: Post-procedure, 1-day, 7-day and 30-day follow up visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
score on a scale | 0 (0)

6. Secondary Outcome: BMSi Scores
Description: BSMi Score is an output measure by the OsteoProbe device to measure bone tissue's resistance to microindentation which can be positively correlated with bone tissue quality.
Time Frame: Procedure
Measure: Mean (Standard Deviation); unit: score
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
score | 77.35 (8.24)

7. Secondary Outcome: Number of Participants With Adverse Events
Description: The number of participants who experienced an adverse event.
Time Frame: Procedure through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
Participants | 1

8. Secondary Outcome: Number of Participants With Device-related Adverse Events
Description: The number of participants who experienced an device-related adverse event.
Time Frame: Procedure through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
Participants | 1

9. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: The number of participants who experienced a Serious adverse event.
Time Frame: Procedure through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
Participants | 0

10. Secondary Outcome: Unanticipated Adverse Device Effects (UADE)
Description: The number of participants who experienced a Unanticipated adverse device effects.
Time Frame: Procedure through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | OsteoProbe System
Number analyzed (Participants) | 40
Participants | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | OsteoProbe System
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsteoProbe System (N=40)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT04628221/Prot_SAP_000.pdf